CLINICAL TRIAL: NCT00112372
Title: A Phase I/IIa, Sequential Cohort, Dose Escalation Trial to Determine the Safety, Tolerability and Maximum Tolerated Dose of AP23573 When Administered Orally in Patients With Refractory or Advanced Malignancies
Brief Title: Study of Oral Ridaforolimus (AP23573, MK-8669) to Treat Patients With Refractory or Advanced Malignancies (MK-8669-016 AM4)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-016; AP23573-05-106
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Cancer
Keywords: unresectable; metastatic; cancer; recurrent; malignancies; progressive
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Recurrence | interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ridaforolimus (Experimental): 10 mg tablet of ridaforolimus administered orally according to one of several different dosing regimens for a four-week treatment cycle.
  Interventions: Drug: Ridaforolimus

INTERVENTIONS:
Drug: Ridaforolimus — 10 mg tablet of ridaforolimus administered orally according to one of several different dosing regimens for a four-week treatment cycle.
  Other Names: AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
The primary objective of this current phase I trial is to study the safety and tolerability of an orally administered dosage form of ridaforolimus. This will be accomplished by an ascending dose study of several dosage regimens in patients with advanced malignancies.

DETAILED DESCRIPTION:
The advent of oral anticancer therapy has created a means to reduce dependency on a system for treating cancer that relies on hospital-based services to administer treatment. While known disadvantages of oral therapies such as potential variable absorption, unpredictable bioavailability and sometimes poor patient compliance pose challenges, the use of orally administered compounds permits investigation of alternative or varied dose regimens, which may ultimately enhance overall patient care.

Ridaforolimus is currently being studied in phase 1 and phase II clinical trials in patients with advanced cancers. Thus far, these trials have demonstrated that ridaforolimus has a favorable safety profile and possesses anticancer activity when administered as a 30-minute intravenous (IV) infusion daily x 5 every-two-weeks or on a weekly schedule. The primary objective of this current phase I trial is to study the safety and tolerability of an orally administered dosage form of ridaforolimus. This will be accomplished by an ascending dose study of several dosage regimens in patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age.
* Patients with a histological/cytological diagnosis of unresectable or metastatic cancer that is refractory to standard therapies or for which no standard therapy exists.
* Patients must must have measurable or nonmeasurable lesions assessable using an appropriate radiographical procedure (e.g., computed tomography (CT) or magnetic resonance imaging (MRI) scans).
* Fertile male or female patients who agree to use approved barrier methods of contraception (non hormonal methods).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Adequate renal and hepatic function, defined as: *Total serum bilirubin ≤ 2 x upper limit of normal (ULN) for the institution; * (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 x ULN for the institution (≤ 5 x if due to hepatic metastases); *Serum albumin ≥ 2 g/dL; Serum creatinine ≤ 2 x ULN for the institution
* Adequate bone marrow function, defined as: * absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; *Platelet count ≥ 100 x 10^9/L
* Serum cholesterol < 350 mg/dL and triglycerides < 400 mg/dL.
* Anticipated life expectancy of ≥ 3 months.
* Able to give and understand a written informed consent.

For the Phase IIa segment, patients must meet the following additional criteria:

* Patients with a histological/cytological diagnosis of metastatic and/or

unresectable sarcoma within one of the following histological subgroups:

* Bone sarcomas
* Leiomyosarcomas
* Liposarcomas

  * Presence of at least one measurable lesion that:
* Can be accurately measured in at least one dimension with longest diameter ≥20 mm using conventional techniques or ≥10 mm with spiral CT scan (or otherwise at least twice the reconstruction interval for CT or MRI scans).
* Previously irradiated lesions may be considered to be measurable provided: 1) there has been documented progression of the lesion(s) since completion of radiotherapy, and 2) the criteria for measurability as outlined above are met.

  * ECOG performance status ≤1

Exclusion Criteria:

* Patients with active central nervous system (CNS) metastases or leptomeningeal disease, not controlled by prior surgery or radiotherapy.
* Prior therapy with rapamycin, rapamycin analogs, or known sensitivity to these agents.
* Prior anticancer treatment, standard or experimental, within 4 weeks prior to the first dose of ridaforolimus (except luteinizing hormone releasing hormone (LH-RH) agonists); the interval is ≥ 2 weeks for signal transduction inhibitors with a half-life known to be < 24 hours, and is ≥ 6 weeks for nitrosourea or mitomycin.
* Concomitant treatment with medications that induce, inhibit, or are

metabolized by cytochrome P450 (CYP3A). Patients should be off these medications 2 weeks prior to the first dose of ridaforolimus.

* Ongoing toxicity associated with prior anticancer therapy (except peripheral neuropathy of ≤ grade 1 by National Cancer Institute (NCI) Terminology Criteria and alopecia).
* Another primary malignancy within the past three years (except in situ carcinoma).
* Known or suspected hypersensitivity to any excipient contained in the study drug.
* Known Grade 3 or 4 hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin).
* Significant uncontrolled cardiovascular disease.
* Active infection requiring systemic therapy.
* Women who are pregnant or lactating.
* Known human immunodeficiency virus (HIV) infection .
* Other life-threatening illness, any medical condition, or organ system dysfunction, which, in the opinion of the Investigator and Sponsor, would either compromise the patient's safety or interfere with evaluation of the safety of ridaforolimus, or could interfere with the absorption of the oral study drug.
* Concurrent treatment with immunosuppressive agents other than prescribed corticosteroids at stable doses for ≥ 2 weeks prior to first planned dose of study drug.
* Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within the last 3 to 4 weeks prior to the first dose of ridaforolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Ridaforolimus When Administered Orally as an Enteric or Film Coated Tablet to Patients With Progressive or Recurrent Malignancies | Cycle 1 (Day 1 to Day 28)
Length of Exposure to Ridaforolimus | Complete duration of study (up to approximately 42 months)
Cumulative Dose of Ridaforolimus | Complete duration of study (up to approximately 42 months)
Number of Participants With Dose Limiting Toxicity (DLT) | Cycle 1 (Day 1 to Day 28)
Efficacy (Clinical Benefit Rate [CBR]) of Ridaforolimus in Advanced Sarcoma | Complete duration of study (up to approximately 42 months)

SECONDARY OUTCOMES:
Area Under the Curve (AUC [0-infinity]) of Ridaforolimus Administered at Different Doses and Regimens | Cycle 1: Days 1 & 15 or 21 (depending on dosing regimen) + Cycle 2 Day 1
Maximum Concentration (Cmax) of Ridaforolimus Administered at Different Doses and Regimens | Cycle 1: Days 1 & 15 or 21 (depending on dosing regimen) + Cycle 2 Day 1
Time at Which Cmax is Reached (Tmax) at Different Doses and Regimens of Ridaforolimus | Cycle 1: Days 1 & 15 or 21 (depending on dosing regimen) + Cycle 2 Day 1
Apparent Terminal Half-Life (t½) of Ridaforolimus | Cycle 1: Days 1 & 15 or 21 (depending on dosing regimen) + Cycle 2 Day 1
Relative Phospho-4E-BP1 (p-4E-BP1) Levels as a Function of Dose | Screening, Cycle 1 Days 1, 2, 11, 15, 16, 22 + Cycle 2 Day 1 or Screening, Cycle 1 Days 1, 2, 11, 21 + Cycle 2 Day 1 (depending on dosing regimen)
Plasma Partitioning | Cycle 1: Days 1 & 15 or 21 (depending on dosing regimen) + Cycle 2 Day 1
Efficacy (Antitumor Activity, as Measured by CBR) of the Study Drug Regimens | Complete duration of study (up to approximately 42 months)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Haluska, M.D., Study Director — Ariad Pharmaceuticals

REFERENCES:
- [Result] Mita MM, Poplin E, Britten CD, Tap WD, Rubin EH, Scott BB, Berk L, Rivera VM, Loewy JW, Dodion P, Haluska F, Sarantopoulos J, Mita A, Tolcher A. Phase I/IIa trial of the mammalian target of rapamycin inhibitor ridaforolimus (AP23573; MK-8669) administered orally in patients with refractory or advanced malignancies and sarcoma. Ann Oncol. 2013 Apr;24(4):1104-11. doi: 10.1093/annonc/mds602. Epub 2012 Dec 4. PMID 23211938
- [Derived] Chawla SP, Staddon AP, Baker LH, Schuetze SM, Tolcher AW, D'Amato GZ, Blay JY, Mita MM, Sankhala KK, Berk L, Rivera VM, Clackson T, Loewy JW, Haluska FG, Demetri GD. Phase II study of the mammalian target of rapamycin inhibitor ridaforolimus in patients with advanced bone and soft tissue sarcomas. J Clin Oncol. 2012 Jan 1;30(1):78-84. doi: 10.1200/JCO.2011.35.6329. Epub 2011 Nov 7. PMID 22067397